CLINICAL TRIAL: NCT02576795
Title: A Phase 1/2, Dose-Escalation, Safety, Tolerability and Efficacy Study of Valoctocogene Roxaparvovec, an Adenovirus-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Patients With Severe Haemophilia A
Brief Title: Gene Therapy Study in Severe Haemophilia A Patients (270-201)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMN 270-201; 2014-003880-38 (EudraCT Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-15 (Estimated); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Severe Haemophilia A
Keywords: Haemophilia A; Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Factor VIII; Coagulants; AAV5 vector
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- valoctocogene roxaparvovec (Experimental): Single administration of valoctocogene roxaparvovec at escalating doses.
  Interventions: Biological: valoctocogene roxaparvovec

INTERVENTIONS:
Biological: valoctocogene roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
  Other Names: BMN 270

SUMMARY:
This study is being conducted by BioMarin Pharmaceutical Inc. as an open label, dose escalation study in order to determine the safety and efficacy of valoctocogene roxaparvovec (an Adenovirus-Associated Virus based gene therapy vector in participants with severe haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Males 18 years or older with established severe Haemophilia A (endogenous FVIII level ≤1 IU/dL) as evidenced by their medical history.
2. Treated/exposed to FVIII concentrates or cryoprecipitate for a minimum of 150 exposure days (EDs)
3. Greater than or equal to 12 bleeding episodes for patients on on-demand FVIII replacement therapy over the previous 12 months. Does not apply to patients on prophylaxis
4. No history of inhibitor, and results from a modified Nijmegen Bethesda assay of less than 0.6 Bethesda Units (BU) 2 consecutive occasions at least one week apart within the past 12 months
5. Sexually active patients must be willing to use an acceptable method of contraception.

Exclusion Criteria:

1. Detectable pre-existing immunity to the AAV5 capsid as measured by adeno-associated virus 5 (AAV5) transduction inhibition (TI) or AAV5 total antibodies
2. Any evidence of immunosuppressive disorder or active chronic infection including hepatis B, hepatitis C, HIV
3. Significant liver dysfunction as defined by abnormal elevation ofliver function tests, or for patients who have undergone liver imaging or biopsy and found to have evidence of grade 3 or higher fibrosis
4. Evidence of any bleeding disorder not related to haemophilia A
5. 12. Treatment with any investigational product within 30 days prior to the end of the screening period, or any previous exposure to any gene transfer therapy
6. Any disease or condition that per the physician's discretion would prevent the patient from fully complying with the requirements of the study including possible corticosteroid treatment outlined in the protocol. The physician may exclude patients unwilling or unable to agree on not using alcohol for the 16-week period following the viral infusion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only
Enrollment: 15 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (5):
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - St. Thomas' Hospital, London
  - The Royal London Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Santos S, Robinson TM, Trueman D. Estimated Long-Term Durability of Valoctocogene Roxaparvovec Treatment in Male patients with Severe Hemophilia A: An Extrapolation of Clinical Data. Adv Ther. 2025 Nov;42(11):5781-5793. doi: 10.1007/s12325-025-03368-4. Epub 2025 Sep 23. PMID 40986187
- [Derived] Symington E, Rangarajan S, Lester W, Madan B, Pierce GF, Raheja P, Millar C, Osmond D, Li M, Robinson TM. Valoctocogene roxaparvovec gene therapy provides durable haemostatic control for up to 7 years for haemophilia A. Haemophilia. 2024 Sep;30(5):1138-1147. doi: 10.1111/hae.15071. Epub 2024 Jul 8. PMID 38975624
- [Derived] Quinn J, Delaney KA, Wong WY, Miesbach W, Bullinger M. Psychometric Validation of the Haemo-QOL-A in Participants with Hemophilia A Treated with Gene Therapy. Patient Relat Outcome Meas. 2022 Jul 18;13:169-180. doi: 10.2147/PROM.S357555. eCollection 2022. PMID 35879931
- [Derived] Fong S, Yates B, Sihn CR, Mattis AN, Mitchell N, Liu S, Russell CB, Kim B, Lawal A, Rangarajan S, Lester W, Bunting S, Pierce GF, Pasi KJ, Wong WY. Interindividual variability in transgene mRNA and protein production following adeno-associated virus gene therapy for hemophilia A. Nat Med. 2022 Apr;28(4):789-797. doi: 10.1038/s41591-022-01751-0. Epub 2022 Apr 11. PMID 35411075
- [Derived] Pasi KJ, Laffan M, Rangarajan S, Robinson TM, Mitchell N, Lester W, Symington E, Madan B, Yang X, Kim B, Pierce GF, Wong WY. Persistence of haemostatic response following gene therapy with valoctocogene roxaparvovec in severe haemophilia A. Haemophilia. 2021 Nov;27(6):947-956. doi: 10.1111/hae.14391. Epub 2021 Aug 11. PMID 34378280
- [Derived] Rosen S, Tiefenbacher S, Robinson M, Huang M, Srimani J, Mackenzie D, Christianson T, Pasi KJ, Rangarajan S, Symington E, Giermasz A, Pierce GF, Kim B, Zoog SJ, Vettermann C. Activity of transgene-produced B-domain-deleted factor VIII in human plasma following AAV5 gene therapy. Blood. 2020 Nov 26;136(22):2524-2534. doi: 10.1182/blood.2020005683. PMID 32915950
- [Derived] Pasi KJ, Rangarajan S, Mitchell N, Lester W, Symington E, Madan B, Laffan M, Russell CB, Li M, Pierce GF, Wong WY. Multiyear Follow-up of AAV5-hFVIII-SQ Gene Therapy for Hemophilia A. N Engl J Med. 2020 Jan 2;382(1):29-40. doi: 10.1056/NEJMoa1908490. PMID 31893514
- [Derived] Rangarajan S, Walsh L, Lester W, Perry D, Madan B, Laffan M, Yu H, Vettermann C, Pierce GF, Wong WY, Pasi KJ. AAV5-Factor VIII Gene Transfer in Severe Hemophilia A. N Engl J Med. 2017 Dec 28;377(26):2519-2530. doi: 10.1056/NEJMoa1708483. Epub 2017 Dec 9. PMID 29224506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites in United Kingdom (Basingstoke, Cambridge, Birmingham, Royal London, London, & Guy's and St. Thomas', London).
Pre-assignment Details: Total of 21 subjects were screened. Of those 21, 6 did not meet the eligibility criteria for enrollment in the study: 5 were found to be adeno-associated virus5 (AAV5) transduction inhibition (TI) or total antibody (TAb) positive, and 1 was assessed as being unable to comply with the requirements of the trial. Fifteen participants were enrolled in 270-201 and received BMN 270 in 1 of 4 dose cohorts
Groups:
- BMN 270 6E12 vg/kg: Cohort 1: 6E12 vector genomes (vg) per kilogram of body weight, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- BMN 270 2E13 vg/kg: Cohort 2: 2E13 vg per kilogram, per kilogram of body weight, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- BMN 270 4E13 vg/kg: Cohort 4: 4E13 vg per kilogram, per kilogram of body weight, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- BMN 270 6E13 vg/kg: Cohort 3: 6E13 vg per kilogram, per kilogram of body weight, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
Period: Overall Study
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Started | 1 | 1 | 6 | 7
Completed | 1 | 1 | 5 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled participants who receive study drug and have at least one Baseline and post-Baseline assessment.
Groups:
- BMN 270 2E13 vg/kg: Cohort 2: 2E13 vg per kilogram, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- BMN 270 4E13 vg/kg: Cohort 4: 4E13 vg per kilogram, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- BMN 270 6E13 vg/kg: Cohort 3: 6E13 vg per kilogram, given as a single intravenous dose (IV)
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
- Total: Total of all reporting groups
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg | Total
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment
  years | 25.0 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 43.0 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 31.3 (9.6) | 30.4 (5.8) | 31.3 (7.8)
Age, Customized [Count of Participants; unit: Participants]
  18 to < 40 years | 1 | 0 | 5 | 6 | 12
  40 to < 60 years | 0 | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 6 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 6 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1 | 2
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 0 | 1 | 5 | 6 | 12
Baseline annualized FVIII usage [Mean (Standard Deviation); unit: IU/kg/year] | 3486.66 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 3022.48 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 4704.16 (2345.75) | 4444.48 (1969.50) | 4389.70 (1965.51)
Baseline annualized number of FVIII infusions [Mean (Standard Deviation); unit: infusions/year] | 87.35 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 103.77 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 142.83 (48.78) | 120.12 (45.94) | 125.93 (45.11)
Baseline ABR (treated bleeds) [Mean (Standard Deviation); unit: bleeds/year] | 2.00 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 3.00 (NA) — The number of participants is 1, so the Standard Deviation was not calculated | 12.17 (15.35) | 17.57 (14.71) | 13.40 (14.26)
Baseline Bleed Counts (treated bleeds) [Count of Participants; unit: Participants]
  0 bleeds/year | 0 | 0 | 1 | 1 | 2
  > 0 to 4 | 1 | 1 | 2 | 1 | 5
  > 4 to 10 | 0 | 0 | 0 | 1 | 1
  > 10 | 0 | 0 | 3 | 4 | 7
History of previous diseases [Count of Participants; unit: Participants] — Some subjects may have multiple conditions.
  In BMN 270-4E13 vg/kg Arm: 4 out of 6 subjects had no history of HepB/HepC/HIV/LD. One subject had multiple conditions (ie Hep B, Hep C and Liver Disease).
  In Total, 10 out of 15 subjects had no history of HepB/HepC/HIV/LD.
  Participants
    Hepatitis B(HepB) | 0 | 0 | 1 | 0 | 1
    Hepatitis C(HepC) | 0 | 1 | 2 | 2 | 5
    Human immunodeficiency virus(HIV) | 0 | 0 | 0 | 0 | 0
    Liver disease(LD) | 0 | 0 | 1 | 0 | 1
Number of target joints [Count of Participants; unit: Participants]
  0 | 0 | 0 | 3 | 1 | 4
  1 | 0 | 0 | 1 | 3 | 4
  2 | 0 | 1 | 0 | 2 | 3
  3 | 1 | 0 | 0 | 0 | 1
  > 3 | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Adverse events (AEs) with onset or worsening after the investigational product were included. Participants with more than one AE of the same category were counted only once for that category.
  Serious adverse event (SAE)
Time Frame: Approximately up to 7 years after dosing
Population: Safety analysis Population: The Safety analysis population was defined as all enrolled participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
Participants
  Participants with any AE | 1 | 1 | 6 | 7
  Participants with any SAE | 1 | 0 | 3 | 5
  Participants with any treatment-related AE | 1 | 0 | 6 | 7
  Treatment-related SAEs | 0 | 0 | 1 | 0
  Participants with any AE of Grade >= 3 | 1 | 1 | 1 | 2
  AEs leading to dose adjustment during infusion | 0 | 0 | 0 | 0
  AEs leading to dose interruption during infusion | 0 | 0 | 0 | 0
  AEs leading to study drug discontinuation | 0 | 0 | 0 | 0
  Participants who died | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participant With Median FVIII Activity Levels >= 5 IU/dL Using Chromogenic Substrate Assay (CSA)
Description: Responder/Non responder status, where a responder was defined as a participant with median FVIII activity of >= 5 IU/dL during Week 13-16 post-BMN 270 infusion
Time Frame: Week 13-16 post-BMN 270 infusion
Population: Full Analysis Set (FAS) population: defined as all enrolled participants who receive study drug and have at least one Baseline and post-Baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
Participants | 0 | 0 | 5 | 7

3. Primary Outcome: Median FVIII Activity as Measured by Chromogenic Substrate Assay During Week 13-16 Post-BMN 270 Infusion
Description: Values for FVIII activity were excluded from analysis if obtained within 72 hours since the last infusion of exogenous FVIII replacement therapy
  FVIII activity levels below the Lower limit of quantitation (LLOQ) will be imputed with 0 IU/dL
  Q1: 25% Percentile; Q3: 75% Percentile
Time Frame: Week 13-16 post-BMN 270 infusion
Population: FAS Population
Measure: Median (Inter-Quartile Range); unit: IU/dL
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
IU/dL | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 16.30 [11.05 to 19.90] | 50.40 [31.30 to 64.95]

4. Secondary Outcome: Annualized Bleeding Rate Requiring Exogenous Factor VIII Replacement Treatment During Week 5 and Beyond
Description: ABR= [Number of bleeding episodes during calculation period] / [Total number of days during the calculation period] ×365.25
  A bleeding episode (treated) was defined as a bleed or symptoms associated with the development of a bleed (or multiple bleeds occurring in the same day) requiring FVIII replacement treatment within 72 hours of the start of the bleed.
  The baseline values for the secondary efficacy endpoints were based on the historical data prior to study enrollment.
  Annualized bleeding rate (ABR)
Time Frame: Week 5 and Beyond (Approximately 7 years post Infusion)
Population: FAS Population
Measure: Mean (Standard Deviation); unit: bleeds/year
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
bleeds/year | 1.87 (NA) — Standard deviation could not be calculated for 1 participant | 6.20 (NA) — Standard deviation could not be calculated for 1 participant | 1.58 (1.97) | 0.75 (1.43)

5. Secondary Outcome: Annualized Factor VIII Utilization During Week 5 and Beyond
Description: Annualized FVIII use (IU/kg/yr.) =[Sum of FVIII use (IU/kg) during calculation period] / [Total number of days during the calculation period] ×365.25
Time Frame: Week 5 and Beyond (Approximately 7 years post Infusion)
Population: FAS Population
Measure: Mean (Standard Deviation); unit: IU/kg/yr
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
IU/kg/yr | 2536.47 (NA) — Standard deviation could not be calculated for 1 participant | 279.27 (NA) — Standard deviation could not be calculated for 1 participant | 331.65 (360.19) | 228.72 (311.68)

6. Secondary Outcome: Annualized Factor VIII Infusion Rate During Week 5 and Beyond
Description: Annualized FVIII infusion rate (count/yr.) = [Number of FVIII replacement infusions during calculation period] / [Total number of days during the calculation period] ×365.25
Time Frame: Week 5 and Beyond (Approximately 7 years post Infusion)
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Infusions/ year
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 1 | 1 | 6 | 7
Infusions/ year | 77.98 (NA) — Standard deviation could not be calculated for 1 participant | 10.09 (NA) — Standard deviation could not be calculated for 1 participant | 10.25 (9.06) | 6.38 (8.19)

ADVERSE EVENTS:
Time Frame: Approximately up to 7 years after dosing
Description: AEs with onset or worsening after the investigational product were included
  Subjects with more than one AE of the same PT were counted only once for that Preferred term (PT)
  AEs were graded for severity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version v4.03
Groups:
- Overall: Overall
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
Arm/Group | BMN 270 6E12 vg/kg | BMN 270 2E13 vg/kg | BMN 270 4E13 vg/kg | BMN 270 6E13 vg/kg | Overall
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/6 | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 3/6 | 5/7 | 9/15
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 6/6 | 7/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 6E12 vg/kg (N=1) | BMN 270 2E13 vg/kg (N=1) | BMN 270 4E13 vg/kg (N=6) | BMN 270 6E13 vg/kg (N=7) | Overall (N=15)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 6E12 vg/kg (N=1) | BMN 270 2E13 vg/kg (N=1) | BMN 270 4E13 vg/kg (N=6) | BMN 270 6E13 vg/kg (N=7) | Overall (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (5)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scleral discolouration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 4 (7) | 6 (11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 5 (8)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 6 (7)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 4 (5)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (3) | 3 (4) | 5 (8) | 10 (16)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 4 (6)
Sputum purulent (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (2) | 2 (3) | 6 (8)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 5 (8) | 7 (9) | 13 (19)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 3 (4) | 9 (10)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coagulation factor VIII level decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coagulation factor VIII level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 5 (9) | 6 (16) | 13 (28)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (1) | 3 (5) | 2 (4) | 7 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 6 (10)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 5 (5) | 6 (8)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (34) | 4 (10) | 8 (45)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 1 (12)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 3 (5)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Sleep deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Typical aura without headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (5) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Idiopathic guttate hypomelanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pregnancy of partner (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT02576795/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02576795/SAP_001.pdf